CLINICAL TRIAL: NCT01066624
Title: A Prospective, Randomized, Comparative Trial of Cryotherapy Versus Caphosol Versus Saline Solution Mouth Washes for the Prevention of Oral Mucositis in Patients With Multiple Myeloma Undergoing Hematopoietic Stem Cell Transplantation.
Brief Title: Comparative Trial of Cryotherapy Versus Caphosol Versus Saline Solution Mouth Washes for the Prevention of Oral Mucositis in Patients With Multiple Myeloma Undergoing Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Juan Toro, Research Fellow, Health Science Specialist, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC20090454H
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Mucositis; Multiple Myeloma
Keywords: Mucositis; Multiple myeloma; Autologous hematopoietic stem cell transplantation
MeSH Terms: conditions — Mucositis; Multiple Myeloma | interventions — Saline Solution; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.9% Sodium Chloride irrigation solution (Active Comparator): Standard of care for prevention and management of oral mucositis (0.9% Sodium Chloride irrigation solution): Patients randomized to this group will be instructed to rinse their mouths twice, with 1 ounce (30 ml) of room temperature 0.9% NaCl (normal saline), 4 times daily after admission and until end of study.
  Interventions: Drug: 0.9% Sodium Chloride irrigation solution
- Cryotherapy (ice chips) (Active Comparator): Patients randomized to this group, on day -2 and -1, will be instructed to place approximately 1 ounce of crushed ice in their mouths 15 minutes prior to the initiation of melphalan infusion. The ice will be allowed to melt and should be replenish as soon as it had completely melted. Patients will be instructed to continue this procedure during the melphalan infusion and for 90 minutes after the end of the infusion. After patients are done with the cryotherapy they will follow the standard of care for prevention and management of oral mucositis until the end of the study.
  Interventions: Other: Cryotherapy (ice chips)
- Calcium phosphate (Caphosol) mouth rinse (Active Comparator): Patients randomized to this group will be instructed to rinse their mouths with Caphosol 4 times daily after admission and until end of study.
  Interventions: Device: Calcium phosphate (Caphosol) Ca2+/PO43- mouth rinse

INTERVENTIONS:
Drug: 0.9% Sodium Chloride irrigation solution — Patients randomized to this group will be instructed to rinse their mouths twice, with 1 ounce (30 ml) of room temperature 0.9% NaCl (normal saline), 4 times daily after admission and until end of study
  Other Names: Normal Saline Solution
  Arms: 0.9% Sodium Chloride irrigation solution
Other: Cryotherapy (ice chips) — Patients randomized to this group, on day -2 and -1, will be instructed to place approximately 1 ounce of crushed ice in their mouths 15 minutes prior to the initiation of melphalan infusion. The ice will be allowed to melt and should be replenish as soon as it had completely melted. Patients will be instructed to continue this procedure during the melphalan infusion and for 90 minutes after the end of the infusion.
  Arms: Cryotherapy (ice chips)
Device: Calcium phosphate (Caphosol) Ca2+/PO43- mouth rinse — Patients randomized to this group will be instructed to rinse their mouths with Caphosol 4 times daily after admission and until end of study.
  Arms: Calcium phosphate (Caphosol) mouth rinse

SUMMARY:
Chemotherapy-induced oral mucositis is the inflammation of the oral mucous membranes, which are tissues that line the mouth. Oral mucositis is caused when chemotherapy attacks and kills the rapidly-dividing cells in the oral mucous membranes. This condition feels like sunburn (or heartburn) on the mucous tissues, and often leads to sores in the mouth or on the tongue. This can cause discomfort, pain, difficulties in eating, and a longer hospital stay. Several therapies appear to either prevent or reduce the severity of mouth ulcers caused by chemotherapy for multiple myeloma. Different strategies are used to try and prevent this condition; a small number of trials found that some of these strategies may be effective. None of the trials had compared head to head the use of saline solution (our standard of care), cryotherapy (ice chips) and Caphosol in patients receiving high-dose melphalan.

The goal of this research study to evaluate the effectiveness of saline solution, cryotherapy, Caphosol for the prevention of oral mucositis in patients with multiple myeloma receiving high-dose chemotherapy followed by autologous hematopoietic stem cell transplantation.

The researchers hope to learn if there are any differences among saline solution, cryotherapy and Caphosol mouth rinse for the prevention of oral mucositis.

DETAILED DESCRIPTION:
INVESTIGATIONAL PLAN Study design This is a single center, prospective, randomized, comparative study to evaluate the effectiveness of saline solution, cryotherapy and Caphosol mouth rinse for the prevention of oral mucositis. Multiple myeloma (MM) patients who are eligible for an autologous hematopoietic stem cell transplantation (HSCT) and are at least 18 years of age will be screened to enroll approximately 165 patients. During the study patients will receive prophylactic fluconazole, acyclovir and antibiotics as appropriate (standard of care). Systemic analgesia will be given for the control of oral pain resulting from mucositis to any of the groups as required. All treatment groups will receive identical oral hygiene care instructions. Treatments not permitted in the study include GM-CSF, palifermin (Kepivance) or other mouthwash and oral coating agents such as Gelclair during the study period to reduce confounding factors.

All patients will receive high-dose melphalan 100 mg /m2/day for 2 days (day -2 and -1) as conditioning regimen followed by autologous HSCT (day 0). After informed consent and completion of screening period, patients will be randomized to any of the three arms. Randomization will be stratified by patient age, sex, and performance status. Patients will be monitored daily post-conditioning until the patients are discharge from the hospital or admitted into an intensive care unit. The oral mucosa will be examined by trained study staff. Oral mucositis will be assessed daily until hospital discharge, after the first day of melphalan, for patients who do not develop oral mucositis or until the oral mucositis resolves for patients who develop any mucositis to a maximum of 30 days. The oral mucositis will be assessed using the World Health Organization (WHO) Mucositis Scale, the Oral Mucositis Assessment Scale (OMAS) and the National Cancer Institute (NCI) Common Toxicity Criteria. At the same time the mucositis-related pain (mouth pain) will be evaluated based on the Wong-Baker Faces Pain Rating Scale and the Numeric Rating Scale (Appendix B). Questionnaire for Patient-reported Oral Mucositis Symptoms (PROMS) Scale will be obtained at screening and every day after first day of melphalan until end of study. All patients will receive the Program's standard oral hygiene instructions prior to initiation of study.

ARM #1:

Standard of care for prevention and management of oral mucositis (0.9% Sodium Chloride irrigation solution): Patients randomized to this group will be instructed to rinse their mouths twice, with 1 ounce (30 ml) of room temperature 0.9% NaCl (normal saline), 4 times daily after admission and until end of study.

ARM #2:

Cryotherapy (ice chips): Patients randomized to this group, on day -2 and -1, will be instructed to place approximately 1 ounce of crushed ice in their mouths 15 minutes prior to the initiation of melphalan infusion. The ice will be allowed to melt and should be replenish as soon as it had completely melted. Patients will be instructed to continue this procedure during the melphalan infusion and for 90 minutes after the end of the infusion. After patients are done with the cryotherapy they will follow the standard of care for prevention and management of oral mucositis until the end of the study.

ARM #3:

Calcium phosphate (Caphosol) Ca2+/PO43- mouth rinse: Patients randomized to this group will be instructed to rinse their mouths with Caphosol 4 times daily after admission and until end of study.

All patients, who develop oral mucositis pain, will follow the Bone Marrow Transplant Program standard of care to control the pain in patients undergoing HDC and autologous HSCT. The Program standard care for oral mucositis pain consists in the use of triple mix solution (lidocaine, Maalox, and diphenhydramine) and analgesics. Patients in the Caphosol rinse arm who develop severe mucositis will be instructed to rinse up to 10 times a day.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria to participate in this study:

* Age 18 years or older
* Patients with diagnosis of MM schedule to receive high-dose melphalan, as a single agent ,for conditioning regimen
* Signed Informed Consent Form

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Patients who have taken palifermin (Kepivance) in the past 90 days
* Patients who have taken any investigational drug in the past 60 days
* Patient who have received radiation therapy in the past 60 days
* Serum creatinine greater than 2 mg/dL
* Patients with mucositis at the time of randomization
* Patients with altered mental status precluding understanding of the informed consent process an/or completion of the necessary assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cesar O Freytes, MD, Study Director — The University of Texas Health Science Center at San Antonio
Locations (1):
- South Texas Veterans Health Care System, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cryotherapy (Ice Chips): Cryotherapy (ice chips): Patients randomized to this group, on day -2 and -1, will be instructed to place approximately 1 ounce of crushed ice in their mouths 15 minutes prior to the initiation of melphalan infusion. The ice will be allowed to melt and should be replenish as soon as it had completely melted. Patients will be instructed to continue this procedure during the melphalan infusion and for 90 minutes after the end of the infusion. After patients are done with the cryotherapy they will follow the standard of care for prevention and management of oral mucositis until the end of the study.
Period: Overall Study
Arm/Group | 0.9% Sodium Chloride Irrigation Solution | Cryotherapy (Ice Chips) | Calcium Phosphate (Caphosol) Mouth Rinse
Started | 38 | 40 | 39
Completed | 38 | 40 | 39
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.9% Sodium Chloride Irrigation Solution | Cryotherapy (Ice Chips) | Calcium Phosphate (Caphosol) Mouth Rinse | Total
Number analyzed (Participants) | 38 | 40 | 39 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 28 | 30 | 88
  >=65 years | 8 | 12 | 9 | 29
Age, Continuous [Mean (Full Range); unit: years] | 61.5 [43 to 70] | 62 [39 to 75] | 62 [45 to 68] | 62 [39 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 36 | 38 | 36 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 5 | 21
  Not Hispanic or Latino | 31 | 31 | 34 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 15 | 11 | 40
  White | 24 | 25 | 28 | 77
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 40 | 39 | 117

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Oral Mucositis
Description: Incidence of grade I-IV oral mucositis
Time Frame: First 30 days post-tranplantation
Measure: Number; unit: percentage of participants
Arm/Group | 0.9% Sodium Chloride Irrigation Solution | Cryotherapy (Ice Chips) | Calcium Phosphate (Caphosol) Mouth Rinse
Number analyzed (Participants) | 38 | 40 | 39
percentage of participants | 66 | 10 | 64

ADVERSE EVENTS:
Arm/Group | 0.9% Sodium Chloride Irrigation Solution | Cryotherapy (Ice Chips) | Calcium Phosphate (Caphosol) Mouth Rinse
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No